CLINICAL TRIAL: NCT04393194
Title: The Effect of Intravaginal Conjugated Estrogen on Ring Pessary Use for Pelvic Organ Prolapse: A Multicenter Randomized, Double- Blind, Placebo Controlled, Clinical Trial
Brief Title: The Effect of Intra-vaginal Conjugated Estrogen Cream on Ring Pessary Use for Pelvic Organ Prolapse
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, zhulan, Director of general gynecology Center, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZS-2164
Record Dates: First submitted 2020-05-10; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Pelvic Floor Prolapse
Keywords: Vaginal estrogen cream
MeSH Terms: interventions — Vaginal Creams, Foams, and Jellies; Dosage Forms; Pessaries

STUDY DESIGN:
Intervention Model Description: Two-arm,Randomized, Double- Blind, Placebo Controlled, Clinical Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal estrogen cream (Experimental): subjects will be treated with the prescribed vaginal medication, 1g per time, q d for the first 2 weeks and then 1g per time, twice a week.
  Interventions: Drug: Vaginal Cream with Applicator [Dose Form]
- vaginal placebo cream (Placebo Comparator): Subjects will be treated with the prescribed vaginal medication, 1g per time, q d for the first 2 weeks and then 1g per time, twice a week.
  Interventions: Drug: Vaginal Cream with Applicator [Dose Form]

INTERVENTIONS:
Drug: Vaginal Cream with Applicator [Dose Form] — Patients with symptomatic POP will be assigned as outpatients. After the initial pessary fitting, the patients will be followed up in 2 weeks. If the prolapse is supported, no discomfort, and the patient decides to continue to use the pessary, the pessary fitting is successful. Patients with successful ring pessary fitting, who agree to participate and sign written consent, will be randomized into the vaginal estrogen group and the placebo group. The patients will be followed up every 3 months after wearing pessary combined with vaginal medication, until 1 year after wearing the pessary.
  Other Names: pessary

SUMMARY:
The primary purpose of this two-arm randomized clinical trial is to determine if in women desiring use of a pessary for pelvic organ prolapse (POP) and are successfully fit, if 1-year use and patient impression of improvement is superior in women using vaginal estrogen cream versus those using a vaginal placebo cream.

DETAILED DESCRIPTION:
The study is a multi-center, randomized trial of women with symptomatic utero-vaginal or post-hysterectomy vaginal vault prolapse desiring non-surgical treatment with a pessary. This study will compare outcomes in women randomized to vaginal estrogen cream or vaginal placebo cream.

Women who meet the inclusion/exclusion criteria will be evaluated. A pessary (ring with support) will be fit by an experienced physician. After successful pessary fitting, they will be randomly divided into experimental active medication and control groups. The experimental group will start intravaginal estrogen cream, and the control group will start intravaginal estrogen-free cream. Then patients will be followed every 3months until 1year.

The purpose of this trial is to evaluate the effect of intravaginal estrogen use on pessary treatment for pelvic organ prolapse, including short-term and long-term use rate, patient impression of improvement, improvement in symptom-specific quality of life and complication incidence.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic POP, stage II, stage III or stage IV
2. Postmenopausal women (patients with serum FSH>40lu/L; or amenorrhea for 12 months)
3. Successfully fit with ring with support pessary
4. Ability to attend the clinical trial and follow-up
5. Patients and their families understand the study, are willing to participate for up to 1 year and can provide written informed consent
6. Willing and able to place vaginal cream

Exclusion Criteria:

1. Acute infection of internal genital tract
2. Hormone replacement therapy in recent 3 months
3. Suspected or untreated lower genital tract tumor
4. Genital fistula
5. Abnormally elevated intra-abdominal pressure (eg ascites, tumor, etc)
6. Life expectancy less than 1 year
7. Vaginal estrogen contraindications, including known or suspected estrogen dependent malignancies (endometrial carcinoma, melanoma), endometrial hyperplasia (thickness of endometrium≥5mm), thrombophlebitis or thromboembolic disease, undiagnosed irregular vaginal bleeding, known or suspected breast cancer, allergy to any component of the estrogen cream and severe liver disease, breast cancer
8. The volume of post-voiding residual is more than 250ml. -

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2020-05-24 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects using the pessary and have very much or much improvement on the patient impression of improvement questionnaire at 1 year between the vaginal estrogen group and the placebo group. | up to 1year after randomization
  1. Sustained wearing with satisfaction: continuous wearing is defined as the use of the pessary after successful fitting test. The continuous wearing time interval is from the start of wearing the pessary to cessation of pessary use.
  2. PGI-I （patient global impression of improvement））is used to evaluate patient impression of improvement. PGI-I is divided into seven levels: very much better, much better, a little bit better, no change, a little bit worse, much worse and very much worse. The patient's response of" very much better" and" much better" is defined as a successful impression of improvement.

SECONDARY OUTCOMES:
1. Comparison of symptom specific distress (PFDI-20) at 6 months and one year in subjects using the pessary in the vaginal estrogen group and the placebo group at 1 year. | up to 1year after randomization
  Questionnaire survey: Relief of symptoms using validated instruments, Pelvic Floor Distress Inventory-20 。PFDI-20 scores 0-300, The higher the score is, the more serious the symptoms of PFD are, the greater the impact on the life of the patients.
1. Comparison of symptom specific impact (PFIQ-7) at 6 months and one year in subjects using the pessary in the vaginal estrogen group and the placebo group at 1 year. | up to 1year after randomization
  Questionnaire survey: Relief of symptoms using validated instruments, pelvic floor impact questionnaire short form 7(PFIQ-7)。PFIQ-7 scores 0-300, the higher the severer negative influence on patient.
1. Comparison of sexual function (PISQ-12) at 6 months and one year in subjects using the pessary in the vaginal estrogen group and the placebo group at 1 year. | up to 1year after randomization
  Questionnaire survey: Relief of symptoms using validated instruments, Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire short form(PISQ-12), PISQ-12 scores 0-48, the higher, the severer negative influence on patient.
Comparison of the adverse events of subjects wearing a pessary in the vaginal estrogen group and the placebo group at 1 year. | up to 1year after randomization
  Complications will be asked and reported during each follow-up

IPD SHARING:
Plan to Share IPD: Yes
Relying on sharing of online database
Supporting Information: CSR
Time Frame: starting 6 months after publication
URL: http://www.chictr.org.cn/index.aspx

REFERENCES:
- [Derived] Zhou Y, Yin R, Zhang Y, Wang X, Jin F, Li X, Peng C, Wang P, Shen H, Weng Q, Xie H, Wang H, Jiang B, Zhou K, Liang N, He Y, Dai Y, Fang Z, Liang S, Zhang Y, Morse A, Zhu L. Effects of intravaginal conjugated oestrogen on pessary continuation for pelvic organ prolapse: multicentre, randomised, double blind, placebo controlled trial. BMJ. 2025 Jun 27;389:e084418. doi: 10.1136/bmj-2025-084418. PMID 40578851
- [Derived] Taithongchai A, Johnson EE, Ismail SI, Barron-Millar E, Kernohan A, Thakar R. Oestrogen therapy for treating pelvic organ prolapse in postmenopausal women. Cochrane Database Syst Rev. 2023 Jul 11;7(7):CD014592. doi: 10.1002/14651858.CD014592.pub2. PMID 37431855